CLINICAL TRIAL: NCT06319144
Title: Effect of Intravenous 5% Dextrose Infusion During Recovery from Anesthesia on the Quality of Early Postoperative Recovery in Patients Undergoing Painless Gastrointestinal Endoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weifang Medical University (Other)
Responsible Party: Principal Investigator, Lin Cheng, Research investigator, Weifang Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: KYLL20240306-1
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Insulin Resistance; Postoperative Nausea and Vomiting; Quality of Recovery; Dizzyness
Keywords: Glucose injection Solution; PONV
MeSH Terms: conditions — Insulin Resistance; Postoperative Nausea and Vomiting; Dizziness | interventions — Glucose; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Active Comparator): Patients in the experimental group were infused intravenously with 5% dextrose (500 ml/h) in the PACU. The study outcomes were collected at three assessment periods, 0-0.5 h, 0.5-6 h, 6-24 h, after anesthesia by an independent investigator.
  Interventions: Other: 5% glucose
- Control group (Active Comparator): Patients in the control group were infused intravenously with 0.9% sodium chloride solution (500 ml/h) in the PACU. The study outcomes were collected at three assessment periods, 0-0.5 h, 0.5-6 h, 6-24 h, after anesthesia by an independent investigator.
  Interventions: Other: 0.9% sodium chloride solution

INTERVENTIONS:
Other: 5% glucose — Patients in the experimental group were infused intravenously with 5% dextrose (500 ml/h) in the PACU.
  Other Names: 5% dextrose; 5% Glucose and sodium chloride injection
  Arms: Experimental group
Other: 0.9% sodium chloride solution — Patients in the control group were infused intravenously with 0.9% sodium chloride solution in the PACU.
  Arms: Control group

SUMMARY:
The aim of this study was to determine the effect of intravenous infusion of 5% dextrose injection during the recovery period of anesthesia for painless gastroenteroscopy on the patient's blood glucose level, incidence of hypoglycemia and time of awakening from anesthesia, postoperative vertigo, postoperative nausea and vomiting, and quality of recovery in the early postoperative period.

ELIGIBILITY:
Inclusion Criteria:

1. patients who meet the indications for painless gastrointestinal endoscopy and are aged 18 to 79 years.
2. The patient or his/her guardian or immediate family members gave informed consent;
3. American Society of Anesthesiology (ASA) anesthesia risk classification ≤ grade III.

Exclusion Criteria:

1. Patients with contraindications to sedation/anesthesia for gastrointestinal endoscopy: e.g., severe hepatic and renal dysfunction, cardiac insufficiency;
2. Patients receiving chemotherapy and opioid treatment; patients with a history of sleep apnea hypoventilation syndrome;
3. Intravenous nutritional support within 8 hours prior to the examination;
4. Patients diagnosed with type I or type II diabetes.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-06-22 (Actual)

PRIMARY OUTCOMES:
Preoperative blood glucose 30min | Measurements taken 0.5 hours Preoperative.
  A fingertip blood glucose concentration of <3.9 mmol/L was used as a diagnostic criterion for hypoglycemia. Severity and incidence of hypoglycemia at 0.5 hours Preoperative.
Postoperative blood glucose 2h | Measured at 2 hours postoperatively.
  A fingertip blood glucose concentration of <3.9 mmol/L was used as a diagnostic criterion for hypoglycemia. Severity and incidence of hypoglycemia at 2 hours postoperatively.
Dizziness level | Approximately 15min after surgery
  The Visual Analogue Scale(VAS) was used to assess the degree of postoperative dizziness in patients undergoing painless gastroenteroscopy.
Dizziness level | Measured at 0.5 hours postoperatively.
  The visual analogue scale (VAS) was used to assess the degree of postoperative dizziness in patients undergoing painless gastroenteroscopy.
Postoperative nausea and vomiting | Measured at 0.5 hours postoperatively.
  The Index of Nausea and Vomiting and Retching (INVR) was used in this study. The scale consists of 8 items with 3 dimensions, which can quantify the number of occurrences, duration and severity of symptoms. The scale is scored using the Likert method, with a total of 32 points on a 5-point scale ranging from 0 to 4. The higher the score, the more severe the symptoms of nausea, vomiting, and dry heaving (entries 1, 6, and 7 are reverse scored). According to the score, nausea, vomiting and dry heaving symptoms can be categorized into five grades: 0, I, II, III and IV, and grade ≥I means that the symptom occurs. The severity and incidence of PONV at 0.5 hours postoperatively.
Postoperative nausea and vomiting | Measured at 2 hours postoperatively.
  The Index of Nausea and Vomiting and Retching (INVR) was used in this study. The scale consists of 8 items with 3 dimensions, which can quantify the number of occurrences, duration and severity of symptoms. The scale is scored using the Likert method, with a total of 32 points on a 5-point scale ranging from 0 to 4. The higher the score, the more severe the symptoms of nausea, vomiting, and dry heaving (entries 1, 6, and 7 are reverse scored). According to the score, nausea, vomiting and dry heaving symptoms can be categorized into five grades: 0, I, II, III and IV, and grade ≥I means that the symptom occurs. The severity and incidence of PONV at 0.5 hours postoperatively.

SECONDARY OUTCOMES:
Anesthesia awakening time | Approximately 30min after surgery
  The clinical routine defines the time of awakening from anesthesia as the time between the cessation of anesthesia administration and the opening of the patient's eyes on call.
Quality of postoperative recovery (QoR40) | Approximately 24hours after surgery
  The QoR-40 scale provides a true and valid reflection of the impact of various factors on the quality of postoperative recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Cheng, B.S, Principal Investigator — Weifang People's Hospital
Locations (1):
- Lin Cheng, Weifang, Shandong, China

IPD SHARING:
Plan to Share IPD: No